CLINICAL TRIAL: NCT01768312
Title: A Multicenter, Randomized, Double-blind Phase Ⅲ Study of Cyclosporine Ophthalmic Soution Group and Cyclosporine Ophthalmic Suspension Group 12 Weeks After Treatment in Moderate to Severe Dry Eye Disease
Brief Title: Study of Cyclosporine Ophthalmic Soution Group and Cyclosporine Ophthalmic Suspension Group
Acronym: Cyclosporine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_TSPR_301
Record Dates: First submitted 2012-12-10; First posted 2013-01-15 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Restasis eye drop (Active Comparator): Cyclosporine 0.05% : 1 drop twice a day for 12 weeks to both eyes
  Interventions: Drug: Cyclosporine ophthalmic solution
- T-sporin eye drop (Experimental): Cyclosporine 0.05% : 1 drop twice a day for 12 weeks to both eyes
  Interventions: Drug: Cyclosporine ophthalmic solution

INTERVENTIONS:
Drug: Cyclosporine ophthalmic solution — 1 drop twice/day for 12 weeks to both eyes
  Other Names: Restasis Eye Drops; Tisporin Eye Drops

SUMMARY:
A Multicenter, Randomized, Double-blind Phase Ⅲ Study of Cyclosporine Ophthalmic Soution Group and Cyclosporine Ophthalmic Suspension Group 12 Weeks After Treatment in Moderate to Severe Dry Eye Disease

DETAILED DESCRIPTION:
The purpose of this clinical Study is Tisporin Eye Drops 0.05%(Cyclosporine ophthalmic solution) group and Restasis Eye Drops 0.05%(Cyclosporine ophthalmic suspension) group 12 weeks after treatment, each treatment group comparisons for evaluation of efficacy and safety in Moderate to Severe Dry Eye Disease.

- Corneal staining test, Ocular surface disease index (OSDI), Tear break up time (TBUT), Non-anesthetic Schirmer test

ELIGIBILITY:
Inclusion Criteria:

* [Patients with moderate-to-severe ocular dry eye]

  1. The sum of corneal fluorescein staining score of 5 or higher (NEI Scale)
  2. Non-anesthetic Schirmer test value ≤ 5mm/5min patients at least one eye score (Non-anesthetic Schirmer test value = 0/5min, nasal stimulation in the same eye, Schirmer test value ≥ 3mm/5min)
  3. Screening both eyes, the corrected visual acuity is 0.2 or more
  4. Despite conventional treatment, the symptoms of dry eye signs (Artificial tear eye drops, sympathetic nervous system stimulant agent, parasympathetic nerve stimulant, etc.)
  5. Negative urine pregnancy test at the screening when women of childbearing age
  6. Medically reliable method of contraception in the case of all women of childbearing age or menopause (1 year after the last menstrual period women) Sterilization (eg, bilateral oophorectomy, hysterectomy) women of childbearing age have not been effective contraception only if you participate in a clinical trial may have been determined to be pregnant by examining whether the voice, maintained during the entire clinical trial period shall that.
  7. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

* 1) Screening visits in the previous 3 months (12 weeks) who participated in the clinical trials of cyclosporine eye drops, or if you used a cyclosporine ophthalmic solutions.

  2) The patients with systemic or ocular disorders affected the test results (ocular surgery, trauma, or disease)
  1. Abnormal eyelid function : Disoders of the eyelids or eyelashes
  2. Ocular allergies or currently under the treatment of allergic diseases of the eye (topical ocular mast cell stabilizer, antihistamine use, etc.)
  3. Cicatricial keratoconjunctivitis caused by herpetic keratopathy, conjunctival scarring (alkali damage, Steven-Johnson syndrome, cicatricial pemphigoid), pterygium, pinguecula, lack of congenital lacrimal, neurogenic keratitis, keratoconus, corneal transplantation 3) current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status 4) The use in clinical trials of drug hypersensitivity reactions in patients 5) patients with contact lens 6) If you use or plan to use punctual plug within 4 weeks 7) Lacrimal punctual occlusion surgery patients 8) Ocular surgery within 3 months (12 weeks) 9) Pregnant women, lactating, or planning to become pregnant 10) The end of the lacrimal gland disease (Nasal stimulation Schirmer test value <3mm/5min) 11) History of malignancy 12) If you are receiving systemic steroids or immunosuppressive treatment 15) In patients with severe renal failure (serum creatinine more than 2.0 times the upper limit of normal) 16) In patients with severe liver dysfunction (ALT or AST of more than 2.0 times the upper limit of normal) 17) Alcohol or drug abuse 18) Pregnant women, lactating women 19) Participating in a Clinical Trial patients who have participated in other clinical trials within three months 20) Patients judged coexisting disease that could interfere with the completion of the treatment or safety of this clinical trial. Patients that other researchers are determined inadequately

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-08-23 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
Corneal staining test | Administered 12 weeks after
  The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source using a yellow filter was evaluated on a 6 point scale according to the oxford grading system

SECONDARY OUTCOMES:
Tear break up time (TBUT) | Administered 4, 8, 12 weeks after
  After blinking blue fluorescein staining of the cobalt blue light source using a yellow filter, it was observed from the blinking point that there was a black spot, a streak pattern or a fluorine defect in the fluorescein-tear layer Was measured in seconds. The measurement results were repeated three times and average values were used.
Corneal staining test | Administered 4, 8 weeks after
  Corneal staining was performed at each visit. The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source using a yellow filter was evaluated on a 6 point scale according to the oxford grading system
Ocular surface disease index (OSDI) | Administered 4, 8, 12 weeks after
  The ocular surface disease index was assessed for ocular surface disease, including visual function (five items), eye symptoms (four items), and environmental factors (three items) , 0 point for no symptoms, 1 point for occasional symptoms, 2 points for symptoms of half a day, 3 points for most symptoms, and 4 points for symptoms during the whole day.
Non-anesthetic Schirmer test | Administered 4, 8, 12 weeks after
  After the eyes were examined, the eyes were wiped and the Schirmer test paper was inserted into the right eye at 1/3 of the lower eyelid without eye anesthesia and inserted into the left eye. After 5 minutes with the eyes closed, the Schirmer test paper was removed from the right side in the order of insertion and the left side removed. The wet length was measured in millimeters and the length of the midpoint was measured when the wet border was oblique.
Conjunctival staining | Administered 4, 8, 12 weeks after
  After lysamine green staining under slit lamps, the conjunctiva was divided into the nasal side and the lateral side, and the degree of nasal conjunctiva and bilateral conjunctival staining was evaluated on a 6-point scale according to the oxford grading system

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of Korea seoul st. Mary's hospital, Seoul, Seocho-Ku, South Korea